CLINICAL TRIAL: NCT06379100
Title: A Randomized, Controlled Clinical Study on Cerebellar ITBS Mode Transcranial Magnetic Stimulation for the Treatment of Alzheimer's Disease
Brief Title: Cerebellar ITBS Mode Transcranial Magnetic Stimulation for the Treatment of Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20232388
Record Dates: First submitted 2024-04-14; First posted 2024-04-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-04

CONDITIONS: Transcranial Magnetic Stimulation; Alzheimer Disease; Magnetic Resonance Imaging; Electroencephalogram
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Alzheimer's disease patients were enrolled by expert neurol ogists who were blinded to treatment allocation. rTMS sessions were performed by dedicated technicians. The Cognitive evaluations and analysis of neuro physiological data were performed by expert neurophysiologists blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Magnetic Stimulation-Real (Experimental): Participants will receive active TMS once daily for four weeks
  Interventions: Device: transcranial magnetic stimulation
- Transcranial Magnetic Stimulation-Sham (Sham Comparator): Participants will receive sham TMS once daily for four weeks
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Intermittent Theta-Burst Transcranial Magnetic Stimulation

SUMMARY:
Study the therapeutic effect and potential neural mechanisms of cerebellar iTBS mode transcranial magnetic stimulation on Alzheimer's disease patients through MRI and EEG.

DETAILED DESCRIPTION:
This study intends to apply intermittent therapy for the first time θ The Outbreak Stimulation (iTBS) mode was used for rTMS treatment in the cerebellum of Alzheimer's disease (AD). This was a randomized, double-blind, parallel, and sham stimulation controlled clinical trial, which included 28 AD patients. All patients were randomly divided into the iTBS group and the sham stimulation group. Collect clinical information, scales, magnetic resonance imaging, TMS synchronous electroencephalography, polysomnography monitoring, etc., and then perform TMS/false stimulation treatment on subjects for 4 weeks (a total of 20 times); After treatment and one month follow-up, relevant scales, magnetic resonance imaging, TMS synchronous electroencephalogram and other data were collected again, and appropriate statistical methods were used to analyze the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 45-80 years old;
2. Meets the NIA-AA standards established by the National Institute on Aging in the United States; Cerebrospinal fluid presents as A β decrease and increase tau protein.

3 The MMSE score ranges from 18 to 26, and the Clinical Dementia Rating (CDR) score is 0.5 to 1 4 At least one adult caregiver 5 patients have received treatment with acetylcholinesterase inhibitors (AChEI) or memantine, such as donepezil, galantamine, or gabalin

* Medication for at least 3 months
* The current dosing regimen remains stable for 8 weeks
* The medication plan remains stable throughout the entire process 6. At least 8 years of educational experience 7 Patients and their families voluntarily sign informed consent forms

Exclusion Criteria:

1. Central nervous system degenerative diseases other than Alzheimer's disease
2. Previous history of epilepsy (excluding febrile seizures in childhood)
3. According to the Diagnostic and Statistical Manual of Mental Disorders, the Fourth Edition - Text Revised Edition (DSM IV-TR) standard meets any of the following:

   * Depression (currently)
   * Schizophrenia
   * Other psychiatric disorders, bipolar disorder, or substance dependence (including alcohol) (within the past 5 years)
4. Cerebrovascular disease (excluding lacunar infarction), severe infection, malignant tumor, accompanied by severe dysfunction of organs such as heart, liver, and kidney
5. There are contraindications for transcranial magnetic stimulation and MRI, or there are metal or implanted devices in the body, such as pacemakers, deep brain stimulators, etc; 6 Use any of the following medications for treatment within the past 3 months:

   * Typical and atypical antipsychotic drugs (such as clozapine, olanzapine)
   * Antiepileptic drugs (such as carbamazepine, topiramate, sodium valproate) 7 has received TMS treatment in the past 8 Participate in clinical trials of any drug within 6 months prior to study registration

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
The changes in CDR（Clinical Dementia Rating） | baseline, 4 weeks after start of the treatment
  The changes in CDR-SB will constitute the major research outcome measure used to assess response to rTMS.There are two scoring methods for the CDR scale, namely Total Score Calculation (CDR-GS) and Sum of Six Content Calculation (CDR-SB). The scoring method used in this study is CDR-SB, with a total score of 18 points. The lower the score, the milder the symptoms

SECONDARY OUTCOMES:
The changes in MMSE(Mini Mental State Examination) | baseline, 4 weeks and 4 weeks after treatment
  The changes in MMSE will constitute the secondary research outcome.The full name of MMSE is mini-mental state examination. The higher the score, the better. In this study, changes in MMSE scores before and after treatment were used as secondary observations.
NPI (Neuropsychiatric Inventory) | baseline, 4 weeks and 4 weeks after treatment
  The changes in NPI will constitute the secondary research outcome. The Neuropsychology Scale (NPI) evaluates 12 neuropsychiatric disorders which included 10 neuropsychiatric symptoms and 2 autonomic neurological symptoms based on the caregiver's perception of the patient's behavior and the perceived distress. The lower the score, the lighter the symptoms.
ADL( Lawton-Brody Activities of Daily Living) | baseline, 4 weeks and 4 weeks after treatment
  The changes in ADL will constitute the secondary research outcome. The ADL evaluates 20 items activities of daily living which included basic life ability and instrument use ability based on the caregiver's perception of the patient's behavior. The lower the score, the lighter the symptoms.
DST (Digital Span Test; Forward and Backward) | baseline, 4 weeks and 4 weeks after treatment
  The changes in DST will constitute the secondary research outcome. Digital span test (DST) was commonly used to evaluate attention ability and instantaneous memory ability.
ADAS-cog（Alzheimer's disease assessment scale) | baseline, 4 weeks and 4 weeks after treatment
  The changes in ADAS-cog will constitute the secondary research outcome. The lower the score, the lighter the symptoms.
DMS(Delayed matching-to-sample task) | baseline, 4 weeks and 4 weeks after treatment
  The DMS paradigm is a commonly used paradigm for studying working memory. This study, combined with EEG monitoring, can investigate the changes in the encoding, maintenance, and retrieval phases of working memory.The changes in DMS will constitute the secondary research outcome.
MEP（Motor evoked potential） | baseline, 4 weeks and 4 weeks after treatment
  MEP is a muscle motor complex potential recorded by stimulating the motor cortex in the contralateral target muscle; Check the overall synchronization and integrity of the transmission and transmission pathways of motor nerves from the cortex to the muscles.The changes in MEP will constitute the secondary research outcome.
MRI measures | baseline, 4 weeks and 4 weeks after treatment
  This study mainly applied resting blood oxygen level dependent functional magnetic resonance imaging (BOLD), arterial spin labeling (ASL), and magnetic resonance diffusion tensor imaging (DTI) techniques to evaluate the changes in functional connectivity of the cerebellar dentate nucleus in healthy subjects and patients before and after 4 weeks of TMS treatment, as well as the changes in the cerebellar cortical white matter fiber bundles one month after treatment.
EEG（electroencephalogram） | baseline, 4 weeks and 4 weeks after treatment
  Use electroencephalography to record resting state electroencephalograms before and after treatment, as well as during follow-up, as well as TMS synchronized electroencephalograms stimulated by single pulse TMS in the bilateral cerebellar dentate nucleus, and task state electroencephalograms during DMS paradigm. Analyzing changes in power spectrum, neural oscillations, and functional connectivity of EEG data before and after treatment and during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, Study Chair — The First Affiliated Hospital of Air Force Medicial University
Locations (1):
- Xijing Hospital of Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xue T, Wu X, Chen S, Yang Y, Yan Z, Song Z, Zhang W, Zhang J, Chen Z, Wang Z. The efficacy and safety of dual orexin receptor antagonists in primary insomnia: A systematic review and network meta-analysis. Sleep Med Rev. 2022 Feb;61:101573. doi: 10.1016/j.smrv.2021.101573. Epub 2021 Nov 26. PMID 34902823
- [Background] GBD 2019 Dementia Forecasting Collaborators. Estimation of the global prevalence of dementia in 2019 and forecasted prevalence in 2050: an analysis for the Global Burden of Disease Study 2019. Lancet Public Health. 2022 Feb;7(2):e105-e125. doi: 10.1016/S2468-2667(21)00249-8. Epub 2022 Jan 6. PMID 34998485
- [Background] Stoodley CJ, Schmahmann JD. Functional topography of the human cerebellum. Handb Clin Neurol. 2018;154:59-70. doi: 10.1016/B978-0-444-63956-1.00004-7. PMID 29903452
- [Background] Stoodley CJ, Schmahmann JD. Functional topography in the human cerebellum: a meta-analysis of neuroimaging studies. Neuroimage. 2009 Jan 15;44(2):489-501. doi: 10.1016/j.neuroimage.2008.08.039. Epub 2008 Sep 16. PMID 18835452
- [Background] Yao Q, Tang F, Wang Y, Yan Y, Dong L, Wang T, Zhu D, Tian M, Lin X, Shi J. Effect of cerebellum stimulation on cognitive recovery in patients with Alzheimer disease: A randomized clinical trial. Brain Stimul. 2022 Jul-Aug;15(4):910-920. doi: 10.1016/j.brs.2022.06.004. Epub 2022 Jun 11. PMID 35700915
- [Background] Beckinghausen J, Sillitoe RV. Insights into cerebellar development and connectivity. Neurosci Lett. 2019 Jan 1;688:2-13. doi: 10.1016/j.neulet.2018.05.013. Epub 2018 May 7. PMID 29746896
- [Background] Marvel CL, Desmond JE. Functional topography of the cerebellum in verbal working memory. Neuropsychol Rev. 2010 Sep;20(3):271-9. doi: 10.1007/s11065-010-9137-7. Epub 2010 Jun 22. PMID 20563894
- [Background] Starowicz-Filip A, Chrobak AA, Moskala M, Krzyzewski RM, Kwinta B, Kwiatkowski S, Milczarek O, Rajtar-Zembaty A, Przewoznik D. The role of the cerebellum in the regulation of language functions. Psychiatr Pol. 2017 Aug 29;51(4):661-671. doi: 10.12740/PP/68547. Epub 2017 Aug 29. English, Polish. PMID 28987056
- [Background] Wu C, Yang L, Feng S, Zhu L, Yang L, Liu TC, Duan R. Therapeutic non-invasive brain treatments in Alzheimer's disease: recent advances and challenges. Inflamm Regen. 2022 Oct 3;42(1):31. doi: 10.1186/s41232-022-00216-8. PMID 36184623
- [Background] Koch G, Casula EP, Bonni S, Borghi I, Assogna M, Minei M, Pellicciari MC, Motta C, D'Acunto A, Porrazzini F, Maiella M, Ferrari C, Caltagirone C, Santarnecchi E, Bozzali M, Martorana A. Precuneus magnetic stimulation for Alzheimer's disease: a randomized, sham-controlled trial. Brain. 2022 Nov 21;145(11):3776-3786. doi: 10.1093/brain/awac285. PMID 36281767
- [Background] Sabbagh M, Sadowsky C, Tousi B, Agronin ME, Alva G, Armon C, Bernick C, Keegan AP, Karantzoulis S, Baror E, Ploznik M, Pascual-Leone A. Effects of a combined transcranial magnetic stimulation (TMS) and cognitive training intervention in patients with Alzheimer's disease. Alzheimers Dement. 2020 Apr;16(4):641-650. doi: 10.1016/j.jalz.2019.08.197. Epub 2020 Jan 16. PMID 31879235
- [Background] Wu X, Ji GJ, Geng Z, Wang L, Yan Y, Wu Y, Xiao G, Gao L, Wei Q, Zhou S, Wei L, Tian Y, Wang K. Accelerated intermittent theta-burst stimulation broadly ameliorates symptoms and cognition in Alzheimer's disease: A randomized controlled trial. Brain Stimul. 2022 Jan-Feb;15(1):35-45. doi: 10.1016/j.brs.2021.11.007. Epub 2021 Nov 6. PMID 34752934
- [Derived] Zhang X, Sun Z, Wu D, Shi X, Song C, Guan X, Hao J, Guo Y, Wang X, Wei D, Liu Z, Zhao J, Jiang W. Effects of cerebellar intermittent theta-burst stimulation on patients with Alzheimer's disease: A randomized controlled trial. J Alzheimers Dis. 2025 Oct;107(3):1187-1199. doi: 10.1177/13872877251366656. Epub 2025 Aug 13. PMID 40801847